CLINICAL TRIAL: NCT03786978
Title: Impact of a Pharmaceutical Care Model in the Reduction of Readmission Rate in Diabetes Melitus Patients in a Public University Hospital, South Brazil
Brief Title: Pharmaceutical Care in the Reduction of Readmission Rates in Diabetes Melitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 150118
Record Dates: First submitted 2018-12-21; First posted 2018-12-26 (Actual); Last update posted 2019-01-07 (Actual); Status verified 2015-09

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes mellitus; Pharmaceutical care; Educational intervention; Pharmacoeconomic evaluation
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial study
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor made a blind evaluation from the study outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Structured pharmaceutical care (Experimental): Patients receive a structured pharmaceutical care until one year after hospital discharge
  Interventions: Behavioral: Structured pharmaceutical care
- Comparator group (Active Comparator): Patient received a single phone call 30 days after basal hospital discharge.
  Interventions: Behavioral: Comparator

INTERVENTIONS:
Behavioral: Structured pharmaceutical care — Patients receive a structured pharmaceutical care from one year after basal hospital discharge
  Arms: Structured pharmaceutical care
Behavioral: Comparator — Patient received a single phone call 30 days after basal hospital discharge.
  Arms: Comparator group

SUMMARY:
Diabetes mellitus (DM) is associated with the frequent use of polypharmacy at different times of administration and requires special attention from the patient or caregivers in order to properly treatment performed. The degree of Functional Literacy in Health is defined as the ability to apply literacy skills to health-related materials, including prescriptions, package inserts, and home care instructions. Several questionnaires are used in research and clinical practice to assess the pronunciation and understanding of commonly used medical terms, as the SAHLPA-18 (Short Assessment of Health Literacy for Portuguese Speaking Adults). The Brief Medication Questionnaire (BMQ) evaluates adherence to medication use from a patient's perspective.

During the basal visit, after the characterization of the sample (n= 100), inpatients from Hospital de Clínicas de Porto Alegre (HCPA) were randomized to interventional or comparator group. The interventional group was follow up during a year after basal discharge. Comparator group received only a phone call, 30 days after the basal discharge, to question how was their healthy status. Readmission rates were evaluated for both groups. Also, a economic evaluation was made to measure the readmission rates in terms of costs.

DETAILED DESCRIPTION:
The first outcome of the clinical study was to measure the readmission rate through a structured pharmaceutical care model after basal hospital discharge and measure the effect of this intervention in terms of readmission reduction in a short term period of 30 days, regardless of the hospitalization reason.

As secondary outcomes the investigators measured the readmission rates after basal hospital discharge and the effect of the intervention in terms of readmission reduction in 60, 90,180 and 365 days after basal hospital discharge. Also, the readmission costs in terms of cost-effectiveness were evaluate.

The sample consisted of 100 patients with DM associated with other comorbidities, hospitalized for any reason in the HCPA, of both sexes, older than 18 years.

Informed consent, demographic and validated questionnaires data were collected in the basal visit. After that, patients were randomized to:

Group 1: comparator; Group 2: structured pharmaceutical intervention.

Seven days after basal hospital discharge, drugs adherence was verified.

The interventional group received pharmaceutical care at basal hospitalization stay, after randomization, have their prescription reviewed until 7 days after discharge of basal hospitalization and also received structured phone calls and mobile SMS (Short Message Service) during one year follow up (30, 60, 180 and 365 days).

Electronic medical records of the included patients (intervention and comparator groups) were reviewed monthly for 12 months, aiming to identify access to emergency services or hospital readmissions at the HCPA and, consequently, the reasons for readmissions and outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with DM and other comorbidities hospitalized for any reason at HCPA
* Patients who are literate or have a literate caregiver;
* Signature in the Term of Consent.

Exclusion Criteria:

* Limited ability to communicate and read in Portuguese and absence of responsible caregiver at the patient room;
* Neuropsychiatric diseases (psychosis, delirium or severe dementia);
* Terminal illness;
* Transplanted patients or users of warfarin, as these patients receive formal guidance from the HCPA pharmaceutical team;
* Auditory or visual impairment that, at the discretion of the investigator, prevents the patient from participating in the study;
* Do not have own mobile number or a close family member living in the same household.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-09-09 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-01-30 (Actual)

PRIMARY OUTCOMES:
Short term readmission rate | 30 days after basal hospital discharge
  Hospital readmissions after basal hospital discharge

SECONDARY OUTCOMES:
Readmission rate - 60 days | 60 days after basal hospital discharge
  Hospital readmissions after basal hospital discharge
Readmission rate - 90 days | 90 days after basal hospital discharge
  Hospital readmissions after basal hospital discharge
Long term readmission rate- 180 days | 180 days after basal hospital discharge
  Hospital readmissions after basal hospital discharge
Long term readmission rate- 365 days | 365 days after basal hospital discharge
  Hospital readmissions after basal hospital discharge
Economic evaluation | 365 days
  Comparison between costs from readmission in both randomized groups

CONTACTS AND LOCATIONS:
Overall Officials: Ticiana C Rodrigues, PhD, Principal Investigator — Federal University of Health Science of Porto Alegre

IPD SHARING:
Plan to Share IPD: No